CLINICAL TRIAL: NCT00990665
Title: Promote Q CRT-D and Quartet Left Ventricular Heart Lead Study
Brief Title: Promote Q Cardiac Resynchronization Therapy Defibrillator (CRT-D) and Quartet Left Ventricular Heart Lead Study
Acronym: Promote Q
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 60024498/E
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: CRT; Heart Failure; LV Leads
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CRT-D and LV lead (Experimental)
  Interventions: Device: CRT-D and LV lead (Quartet™ lead and Promote Q® device system)

INTERVENTIONS:
Device: CRT-D and LV lead (Quartet™ lead and Promote Q® device system) — Promote Q CRT-D and Quartet LV lead

SUMMARY:
The objective of this study is to assess the safety and efficacy of the Quartet™ lead and Promote Q® device system in a patient population indicated for cardiac resynchronization therapy.

ELIGIBILITY:
Inclusion Criteria:

* Approved indication per ACC/AHA/HRS guidelines for implantation of a CRT-D system for treatment of heart failure or lifethreatening ventricular tachyarrhythmia(s)
* Receiving a new implant or undergoing an upgrade from an existing ICD or pacemaker implant with no prior LV lead placement.
* Ability to provide informed consent for study participation and is willing and able to comply with the prescribed follow-up tests and schedule of evaluations

Exclusion Criteria:

* Have had a recent CVA or TIA within three months of enrollment
* Have a contraindication for an emergency thoracotomy
* Have a hypersensitivity to a single 1.0mg dose of dexamethasone sodium phosphate or short term contact with heparin
* Have a classification of Status 1 for cardiac transplantation or consideration for transplantation over the next 3 months
* Have undergone a cardiac transplantation within 40 days of enrollment
* Have had a recent myocardial infarction, unstable angina or cardiac revascularization (PTCA, Stent or CABG) within 40 days of enrollment
* Are currently participating in a clinical investigation that includes an active treatment arm
* Are pregnant or planning to become pregnant during the duration of the study
* Have a life expectancy of less than 6 months due to any condition
* Are less than 18 years of age
* Are unable to comply with the follow up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gery Tomassoni, MD, Study Chair — Central Baptist Hospital
Locations (24):
- United States (24):
  - University Hospital of Alabama at Birmingham, Birmingham, Alabama
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Glendale Memorial Medical Center, Glendale, California
  - University of Southern California, Los Angeles, California
  - ACS Research Group, Mountain View, California
  - Regional Cardiology Associates, Sacramento, California
  - Scripps Green Hospital, San Diego, California
  - Orlando Heart Center, Orlando, Florida
  - The Heart and Vascular Institute of Florida - S. Pinellas, St. Petersburg, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Midwest Heart Foundation, Lombard, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - Lahey Clinical Medical Center, Burlington, Massachusetts
  - Thoracic Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Mount Sinai Hospital, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - EMH Regional Medical Center, Elyria, Ohio
  - Lancaster Heart Foundation, Lancaster, Pennsylvania
  - Methodist University Hospital, Memphis, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - Arrhythmia Center for Southern Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Tomassoni G, Baker J, Corbisiero R, Love C, Martin D, Niazi I, Sheppard R, Worley S, Beau S, Greer GS, Aryana A, Cao M, Harbert N, Zhang S; Promote(R) Q CRT-D and Quartet(R) Left Ventricular Heart Lead Study Group. Postoperative performance of the Quartet(R) left ventricular heart lead. J Cardiovasc Electrophysiol. 2013 Apr;24(4):449-56. doi: 10.1111/jce.12065. Epub 2013 Jan 22. PMID 23339555

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CRT-D and LV Lead
Started | 178
Completed | 130
Not Completed | 48
Not completed — Unsuccessful Implant | 8
Not completed — Death | 29
Not completed — Heart Transplant | 1
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 1
Not completed — System Explant | 3

BASELINE CHARACTERISTICS:
Arm/Group | CRT-D and LV Lead
Number analyzed (Participants) | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 140
  More than one race | 2
  Unknown or Not Reported | 2
New York Heart Association Class [Number; unit: participants] — The New York Heart Association (NYHA) classification system is the most commonly used classification system for heart failure. Class I (least severe): No symptoms and no limitations on ordinary physical activity; Class II: Mild symptoms and slight limitations on ordinary physical activity; Class III: Marked limitation on activity due to symptoms; Class IV (most severe): Severe limitations and even symptoms at rest.
  participants
    Class III | 175
    Class IV | 3

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Left Ventricular Lead-Related Complications Through 3 Months
Description: The primary safety endpoint for this study is freedom from left ventricular lead-related complications through 3 months.
Time Frame: 3 months
Population: Patients implanted with a Promote Q CRT-D device and Quartet LV lead.
Measure: Number (97.5% Confidence Interval); unit: percentage probability
Arm/Group | CRT-D and LV Lead
Number analyzed (Participants) | 178
percentage probability | 96 [93 to NA] — Upper bound was not calculated for this outcome measure with one sided hypothesis

2. Primary Outcome: Freedom From System-related Complications Through 3 Months
Description: The co-primary safety endpoint for this study is freedom from system-related complications through 3 months.
Time Frame: 3 Months
Population: Participants implanted with a Promote Q CRT-D device and Quartet LV lead.
Measure: Number (97.5% Confidence Interval); unit: percentage probability
Arm/Group | CRT-D and LV Lead
Number analyzed (Participants) | 178
percentage probability | 92 [88 to NA] — Upper bound was not calculated for this outcome measure with one sided hypothesis

3. Primary Outcome: The Primary Effectiveness Endpoint for the Promote Q System Was the Responder Rate to Biventricular Pacing at 3 Months.
Description: The primary effectiveness endpoint for the Promote Q system was the responder rate to biventricular pacing at 3 months. A responder per protocol was defined as a patient with an LV pacing threshold of <2.5 V at 0.5ms in the D1-M2 pacing configuration (Vector 1) AND at least one other non-standard programmable biventricular lead vector. Non-standard vectors included Vector 2 (D1-P4), Vector 4 (M2-P4), Vector 6 (M3-M2), Vector 7 (M3-P4), Vector 8 (M3-RV coil), Vector 9 (P4-M2) and Vector 10 (P4-RV coil).
Time Frame: 3 Months
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Groups:
- Patients Per Statistical Analysis Plan: Total number of participants enrolled in the study (with an attempted implant of a Promote Q CRT-D and Quartet LV lead including unsuccessful implants).
- Patients Per Complete Case Analysis: Complete case analysis includes only the number of patients that were successfully implanted with the Promote Q CRT-D and Quartet LV lead.
Arm/Group | Patients Per Statistical Analysis Plan | Patients Per Complete Case Analysis
Number analyzed (Participants) | 178 | 162
percentage of participants | 79.2 [72.5 to NA] — Upper bound was not calculated for this outcome measure with one sided hypothesis | 83.3 [76.7 to NA] — Upper bound was not calculated for this outcome measure with one sided hypothesis

ADVERSE EVENTS:
Groups:
- CRT-D and LV Lead: CRT-D and LV Lead
Arm/Group | CRT-D and LV Lead
Serious Adverse Events (participants affected / at risk) | 0/178
Other Adverse Events (participants affected / at risk) | 76/178
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT-D and LV Lead (N=178)
Complications (Cardiac disorders) | 28 (36)
Observations (Cardiac disorders) | 48 (59)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No